CLINICAL TRIAL: NCT02273219
Title: Phase Ib Trial of AEB071, a PKC Inhibitor, in Combination With BYL719, a PI3Kα Inhibitor, in Patients With Metastatic Uveal Melanoma
Brief Title: Trial of AEB071 in Combination With BYL719 in Patients With Melanoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Columbia University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: AAAN4901; CAEB071AUS01T (Other: Novartis)
Record Dates: First submitted 2014-10-17; First posted 2014-10-23 (Estimated); Last update posted 2023-08-15 (Actual); Status verified 2023-08

CONDITIONS: Uveal Melanoma
Keywords: Uveal; Melanoma; Advanced uveal melanoma
MeSH Terms: conditions — Uveal Melanoma; Melanoma | interventions — sotrastaurin; Alpelisib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Dose 1: AEB071 and BYL719 (Experimental): AEB071, oral, 100 mg twice daily BYL719, oral, 200 mg daily
  Interventions: Drug: AEB071; Drug: BYL719
- Dose 2: AEB071 and BYL719 (Experimental): AEB071, oral, 200 mg twice daily BYL719, oral, 250 mg daily
  Interventions: Drug: AEB071; Drug: BYL719
- Dose 3: AEB071 and BYL719 (Experimental): AEB071, oral, 200 mg twice daily BYL719, oral, 300 mg daily
  Interventions: Drug: AEB071; Drug: BYL719
- Dose 4: AEB071 and BYL719 (Experimental): AEB071, oral, 200 mg twice daily BYL719, oral, 350 mg daily
  Interventions: Drug: AEB071; Drug: BYL719
- Dose 5: AEB071 and BYL719 (Experimental): AEB071, oral, 300 mg twice daily BYL719, oral, 350 mg daily
  Interventions: Drug: AEB071; Drug: BYL719

INTERVENTIONS:
Drug: AEB071 — Oral, 100-400 mg twice daily A potent, oral, selective inhibitor of the classical Protein Kinase C (PKC)
  Other Names: Sotrastaurin
Drug: BYL719 — Oral, 200-350 mg daily An oral class I α-specific PI3K inhibitor belonging to the 2-aminothiazole class of compounds
  Other Names: NVP-BYL719

SUMMARY:
Primary objective is to define the maximum tolerated dose (MTD) for the combination of AEB071 and BYL719. Secondary objectives are to define the safety and tolerability of AEB071 and BYL719.

DETAILED DESCRIPTION:
Uveal melanoma is the most common primary intraocular malignancy in adults and is thought to be particularly resistant to systemic treatment, and no systemic therapy has yet been demonstrated to improve survival. Drugs commonly used to treat advanced cutaneous melanoma rarely achieve durable responses in patients with uveal melanoma. Because of the lack of effective systemic treatment options, outcomes are poor once metastatic disease occurs, and the median survival from the time of the development of distant metastatic disease is 6 to 12 months. Although it is clear that novel effective therapies are desperately needed for this disease, the development of such therapies has been hampered by the rarity of uveal melanoma.

ELIGIBILITY:
Inclusion Criteria:

* Metastatic histologically or cytologically confirmed uveal melanoma with pathologic confirmation at a participating center that is judged to be progressive in the opinion of the treating physician.
* Measurable disease. Patients with biopsy-proven metastatic disease that do not meet criteria for measurable disease may be eligible at the discretion of the principal investigator.
* Prior cytotoxic therapy and immunotherapy are allowed. For the dose escalation, prior targeted therapy with a MEK inhibitor, Protein Kinase C inhibitor, Akt, or mechanistic target of rapamycin (mTOR) inhibitor are allowed. For the dose expansion cohort, no prior PKC, Akt, or mTOR inhibitors are allowed. Local therapies such as radiofrequency ablation or cryotherapy for metastatic disease are permitted but must have been performed at least 21 days prior to initiation of study therapy.
* Age greater than or equal to 18 years
* Willingness to undergo core biopsies at baseline, mid-Cycle 1, and/or at progression unless contraindicated by medical risk in the opinion of the treating physician.
* Easter Cooperative Oncology Group (ECOG) performance status less than or equal to 2 (Karnofsky greater than or equal to 60 percent).
* Life expectancy of greater than 3 months.
* Able to swallow and retain medication and does not have any clinically significant gastrointestinal abnormalities that may alter absorption such as malabsorption syndrome or major resection of the stomach or bowels.
* Fasting plasma glucose (FPG) less than 140 mg/dL / 7.8 mmol/L.
* All prior treatment-related toxicities must be grade less than or equal to 1 (except alopecia).
* Patients must have adequate organ and marrow function within 14 days of starting Cycle 1, Day 1 of therapy
* Women of child-bearing potential and men must agree to use adequate contraception prior to study entry and for the duration of study participation. Women of child-bearing potential must have a negative serum pregnancy test within 14 days prior to registration.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* History of another malignancy except for those who have been disease-free for 24 months. Patients with a history of completely resected non-melanoma skin cancer and/or patients with indolent secondary malignancies not requiring active therapy are eligible.
* Any major surgery or extensive radiotherapy within 28 days prior to screening
* Use of other investigational drugs within 28 days (or five half-lives, whichever is longer) preceding the first dose of AEB071 and BYL719.
* Symptomatic or untreated leptomeningeal or brain metastases or spinal cord compression. Treated brain metastases must have been stable for at least 1 month.
* Have a known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to AEB071 or BYL719.
* Current use of a prohibited medication.
* Type I Diabetes Mellitus (DM), Type II DM patients requiring insulin for chronic blood glucose control, and any patients with a fasting blood glucose greater than 140 mg/dL at screening.
* History or evidence of cardiovascular risk.
* Known Human Immunodeficiency Virus (HIV), Hepatitis B Virus (HBV), or Hepatitis C Virus (HCV) infection (with the exception of chronic or cleared HBV and HCV infection, which will be allowed).
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection and psychiatric illness/social situations that would limit compliance with study requirements.
* Patients with impairment of gastrointestinal function or gastrointestinal disease that could interfere with the absorption of AEB071 or BYL719 (e.g. ulcerative disease, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, or small bowel resection).
* Patients who have received prior systemic anti-cancer treatment, such as cyclical chemotherapy or biological therapy within a period of time that is shorter than the cycle length used for that treatment (e.g. 6 weeks for nitrosourea, mitomycin-C) prior to starting study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-11-19 (Actual); Primary Completion 2017-10-18 (Actual); Study Completion 2018-07-02 (Actual)

PRIMARY OUTCOMES:
Total maximum tolerated dose (in milligrams) of AEB071 in combination with BYL719 | 4 years (approximately)
  Establish the maximum tolerated dose (up to 400 mg twice daily) for AEB071 and up to 350 mg daily for BYL719

SECONDARY OUTCOMES:
Number of participants with adverse events | 4 years (approximately)
  Obtain safety data of the combination therapy of AEB071 with BYL719
Change in area under the curve (AUC) for the combination of AEB071 and BYL719 | Cycle 1 Day 1, pre-dose, .5, 1, 2, 4, 6, 8, and 24 hours post dose, Cycle 1, Day 8, pre-dose, .5, 1, 2, 4, 6, and 8 hours post dose, Cycle 1 Day 15, pre-dose, Cycle 2-3-4-5-6 Day 1, pre-dose
  To evaluate the pharmacokinetic properties of the combination of AEB071 and BYL719 at varying dose levels utilizing standard pharmacokinetic parameters such as peak concentration (Cmax) and area under the curve (AUC) of AEB071 and BYL719 in plasma samples.
Change in peak concentration (Cmax) for the combination of AEB071 and BYL719 | Cycle 1 Day 1, pre-dose, .5, 1, 2, 4, 6, 8, and 24 hours post dose, Cycle 1, Day 8, pre-dose, .5, 1, 2, 4, 6, and 8 hours post dose, Cycle 1 Day 15, pre-dose, Cycle 2-3-4-5-6 Day 1, pre-dose
  To evaluate the pharmacokinetic properties of the combination of AEB071 and BYL719 at varying dose levels utilizing standard pharmacokinetic parameters such as peak concentration (Cmax) and area under the curve (AUC) of AEB071 and BYL719 in plasma samples.
Number participants who respond to therapy | 4 years (approximately)
  Clinical benefit rate will be assessed as overall object response rate, using metric measurements on imaging scans.
Change in numerically calculated toxicity burden (0-10) | baseline, Cycle 1 Day 8, Day 15, and Day 22, Cycle 2 and above, End of Treatment, 28 day Follow-Up visit
  To explore the toxicity burden on the patient during treatment as perceived by the patient and the physician.
Mean months of overall survival | 4 years (approximately)
  Overall survival will be calculated in months, starting at time of enrollment.

CONTACTS AND LOCATIONS:
Overall Officials: Richard Carvajal, MD, Principal Investigator — Columbia University
Locations (3):
- United States (3):
  - Bascom Palmer Eye Institute of University Of Miami Medical Center, Miami, Florida
  - Columbia University Medical Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York

IPD SHARING:
Plan to Share IPD: Undecided